CLINICAL TRIAL: NCT00702117
Title: Ajmaline Utilization in the Diagnosis and Treatment of Cardiac Arrhythmias
Acronym: AJUAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: José Brugada, Hospital Clinic de Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AJUAR; EudraCT number:2007-006334-33
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-01

CONDITIONS: Atrial Fibrillation; Tachycardia, Ventricular; Brugada Syndrome
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia, Ventricular; Brugada Syndrome | interventions — Flecainide; Ajmaline; Procainamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- A (Active Comparator): IV flecainide in atrial fibrillation
  Interventions: Drug: flecainide
- B (Experimental): IV ajmaline in atrial fibrillation
  Interventions: Drug: ajmaline
- c (Active Comparator): iv procainamide in ventricular tachycardia
  Interventions: Drug: procainamide
- d (Experimental): iv ajmaline in ventricular tachycardia
  Interventions: Drug: ajmaline
- e (Active Comparator): iv flecainide in diagnosis of Brugada Sd
  Interventions: Drug: flecainide
- f (Experimental): iv ajmaline in diagnosis of Brugada Sd
  Interventions: Drug: ajmaline

INTERVENTIONS:
Drug: flecainide — 2 mg/kg iv in 10 minutes
  Arms: A; e
Drug: ajmaline — 1 mg/kg iv in 10 minutes
  Arms: B; d; f
Drug: procainamide — 10 mg/kg iv in 10 minutes
  Arms: c

SUMMARY:
The study evaluates 3 different populations:

It is an open, randomized, parallel-group study comparing the effectiveness of intravenous (iv) ajmaline with currently used antiarrhythmic drugs in the acute treatment of :

1. recent-onset atrial fibrillation versus iv flecainide
2. sustained monomorphous ventricular tachycardia versus iv procainamide

The study also evaluates in an open, randomized, crossover study, the use of iv ajmaline versus iv flecainide in the diagnosis of Brugada syndrome

ELIGIBILITY:
Inclusion Criteria:

* AF: Patients with isolated, idiopathic, sustained, symptomatic, recent onset(>10 minutes to <24 hours) atrial fibrillation.
* VT: Patients with ventricular tachycardia with good haemodynamic tolerability attending the emergency room or induced at the electrophysiology lab during testing for ventricular arrhythmias.
* Brugada Sd (BrS): First-degree relatives of a patient with Brugada Syndrome with a ECG non-diagnostic of the BrS.

Exclusion Criteria:

* General: Pregnancy
* AF: Pre-existing heart disease.
* Secondary AF
* 2nd and 3rd degree AV block or RBBB associated with LAFB or LPFB (bifascicular block).
* LVF<40%.
* Moderate-severe liver failure.
* AF with haemodynamic compromise.
* VT:VT with haemodynamic compromise.
* BrS:Pre-existing heart disease.
* 2nd and 3rd degree AV block or RBBB associated with LAFB or LPFB (bifascicular block).
* Moderate-severe liver failure.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with reversion of atrial fibrillation | 1 hour
Proportion of patients with reversion of ventricular tachycardia | 15 min
Proportion of subjects developing EKG pattern diagnostic of Brugada Sd. after provocation test. | 1 hour

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Servicio de Cardiología, Hospital Clínic, Barcelona, Barcelona
  - Hospital Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital Puerta de Hierro, Madrid, Madrid
  - Hospital La Fe, Valencia, Valencia